CLINICAL TRIAL: NCT01936831
Title: The Early Bactericidal Activity of High-Dose or Standard-Dose Isoniazid Among Adult Participants With Isoniazid-Resistant or Drug-Sensitive Tuberculosis
Brief Title: High-Dose Isoniazid Among Adult Patients With Different Genetic Variants of INH-Resistant Tuberculosis (TB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5312; UM1AI068636 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: 5mg Cohort (Experimental): Group 1 participants had an M. tuberculosis strain with an inhA mutation only. 5 mg cohort received Isoniazid 5 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
  Interventions: Drug: Isoniazid; Dietary Supplement: Vitamin B6
- Group 1: 10mg Cohort (Experimental): Group 1 participants had an M. tuberculosis strain with an inhA mutation only. 10 mg cohort received Isoniazid 10 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
  Interventions: Drug: Isoniazid; Dietary Supplement: Vitamin B6
- Group 1: 15mg Cohort (Experimental): Group 1 participants had an M. tuberculosis strain with an inhA mutation only. 15 mg cohort received Isoniazid 15 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
  Interventions: Drug: Isoniazid; Dietary Supplement: Vitamin B6
- Group 2: 5mg Cohort (Active Comparator): Group 2 participants had an M. tuberculosis strain with neither inhA nor katG mutations. All Group 2 participants received Isoniazid 5 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
  Interventions: Drug: Isoniazid; Dietary Supplement: Vitamin B6
- Group 3: 15mg Cohort (Experimental): Group 3 participants had an M. tuberculosis strain with a katG mutation with or without an inhA mutation. 15mg cohort received Isoniazid 15 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
  Interventions: Drug: Isoniazid; Dietary Supplement: Vitamin B6
- Group 3: 20mg Cohort (Experimental): Group 3 participants had an M. tuberculosis strain with a katG mutation with or without an inhA mutation. 20mg cohort received Isoniazid 20 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
  Interventions: Drug: Isoniazid; Dietary Supplement: Vitamin B6

INTERVENTIONS:
Drug: Isoniazid — INH was available in 100 mg tablets. INH was administered orally daily in the morning on an empty stomach. Doses of INH were given according to the weight bands and by cohort.
  Other Names: INH
Dietary Supplement: Vitamin B6 — Vitamin B6 was administered at >= 25 mg daily and was obtained locally for use by study participants.

SUMMARY:
Isoniazid (INH) is a drug commonly used to treat tuberculosis (TB) worldwide. Sometimes, the bacteria that cause TB can become resistant to INH. Resistance means that bacteria have adapted to a drug and are able to live in the presence of the drug. When TB becomes resistant to INH, INH does not work as well at fighting the bacteria. This study treated people with INH-resistant TB with different doses of INH to see if INH can still fight the bacteria if the dose is increased. We evaluated how well the drug works at higher doses for participants who have resistant TB as well as how well the drug works at regular doses for participants who have TB that is not resistant. The study also evaluated the safety and tolerability of the different doses of INH. Tolerability is how well people can put up with the side effects of a drug. Using increased doses of INH to treat TB that is resistant to INH is experimental and has not been approved by regulatory authorities. While there is some evidence that this approach will work, this has not yet been proven.

DETAILED DESCRIPTION:
A5312 was a two-stage, two-step, phase IIa, open-label, randomized clinical trial among adult participants with sputum smear positive pulmonary TB evaluating the early bacterial activity (EBA).

No study drug was administered under Step 1. Data collected in Step 1: (a) determined eligibility to Step 2, and (b) allowed characterization of INH MICs in three groups. Groups 1, 2, and 3 consist of participants infected with TB with inhA mutations, with drug susceptible TB (DS-TB), and with TB with katG resistance-conferring mutations, respectively.

Participants enrolled to Step 2 received the study drug, INH, which was given with vitamin B6 >=25 mg daily, by mouth. During both stages, participants in Group 1 who met Step 2 entry criteria were randomized to receive 5, 10, or 15 mg/kg of INH daily for 7 days. During Stage 2, participants in Group 2 who met Step 2 entry criteria received 5 mg/kg of INH daily for 7 days. Under protocol version 3.0 during Stage 2, participants in Group 3 who met Step 2 entry criteria were randomized to receive 15 or 20 mg/kg of INH daily for 7 days. After completion of 7 days of INH alone, participants were referred to begin standard anti-TB chemotherapy according to local guidelines.

In Step 2, prior to initiation of treatment, sputum was collected for quantitative culture on solid medium (for colony forming units (CFU) for Groups 1 and 2 only) and liquid medium (for determination of time to positivity (TTP) for all groups). Sixteen-hour sputum collections were performed daily during INH treatment, as per standard early bacterial activity (EBA) methodology. Sampling for PK analysis was performed at steady state on Day 6 (±1). Safety and tolerability were monitored via clinical evaluations throughout the study and through scheduled laboratory evaluations.

The study consisted of two stages, as follows:

Stage 1-Pilot study to ensure feasibility:

The goal of Stage 1 was to demonstrate feasibility, not treatment efficacy.

Participants were recruited at a single clinical site. All eligible participants entered Step 1 of the study (determination of INH resistance, measurement of INH minimum inhibitory concentrations (MIC)). Among Group 1 participants who met the Step 2 entry criteria, 15 participants were randomized 1:1:1 to receive 5, 10, or 15 mg/kg daily of INH for 7 days with evaluations performed as described above.

Stage 1 completed March 26, 2015. A total of 15 Group 1, 44 Group 2, and 12 Group 3 participants were enrolled in Step 1 only during Stage 1. These participants did not receive study treatment. They provided sputum samples for MIC determination.

Stage 2-Main study:

During Stage 2, Group 1 participants who met Step 2 entry criteria were randomized 1:1:1 to receive 5, 10, or 15 mg/kg of INH daily for 7 days. Group 2 participants who met Step 2 entry criteria were enrolled and received INH at a dose of 5 mg/kg daily. Group 3 participants who met Step 2 entry criteria were enrolled and randomized 1:1 to receive INH at a dose of 15 or 20 mg/kg daily.

In Stage 1, Group 1 participants who did not meet Step 2 entry criteria, all Group 2 participants and all Group 3 participants were referred to a local TB program for treatment. In Stage 2, Group 1, 2 and 3 participants who did not meet Step 2 entry criteria, were referred to a local TB program for treatment.

Protocol Versions:

Key differences in protocol versions include the following:

* Study entry criteria were changed from protocol versions 1.0 to 2.0

  * No longer excluded individuals for antiretroviral therapy use
  * Exclusion of individuals with any MDR-TB treatment with second-line anti-TB drugs was relaxed to exclude only those with more than 7 cumulative days of use.
* Protocol version 2.0 allowed additional sites to enroll participants.
* Under protocol versions 1.0 and 2.0, eligible individuals in Group 1 and Group 2 could enroll in Step 1 and Step 2, and eligible individuals in Group 3 could be enrolled in Step 1 only. Under protocol version 3.0, eligible individuals in Group 3 could enroll in Step 1 and Step 2.
* Early bactericidal activity was described using both solid culture CFU and liquid culture TTP under protocol versions 1.0 and 2.0. Under protocol version 3.0, early bactericidal activity was measured by liquid culture TTP only.
* There were technical difficulties with measuring the isoniazid minimum inhibitory concentration using 1% agar solution for participants enrolled under protocols versions 1.0 and 2.0. For protocol version 3.0, the Thermo Fisher MYCOTB Sensititre plate was substituted to overcome the technical difficulties.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* New or recurrent pulmonary TB with sputum positive for acid-fast bacilli on direct microscopy of at least grade 1+ (International Union Against Tuberculosis and Lung Disease [IUATLD] scale) at the study laboratory on at least one pre-treatment sputum sample within 14 days prior to entry.
* Infected with an M. tuberculosis strain for which Hain GenoType MTBDRplus genotype, performed at the study laboratory within 14 days prior to study entry, reveals one of the following results for INH susceptibility testing:

  * inhA promoter or functional mutation only (Group 1 participants, eligible for Steps 1 and 2)
  * No mutations in the inhA or katG genes (Group 2 participants, eligible for Step 1 and, during Stage 2 of the study, also eligible for Step 2)
  * katG mutation with or without an inhA mutation (Group 3 participants, eligible for Step 1 and, during Stage 2 of the study, also eligible for Step 2)
* Ability and willingness of the participant or legal guardian/representative to provide informed consent.

Inclusion Criteria for Step 2:

* Entry into Step 1.
* During Stage 1 of the protocol: inhA promoter or functional mutation only (Group 1).
* During Stage 2 of the protocol: inhA promoter or functional mutation only (Group 1) OR mutations in neither inhA nor katG genes (Group 2) or mutation in the katG gene, with or without mutations in inhA promoter or functional genes (Group 3).
* Body weight: 40 kg to 90 kg, inclusive.
* Laboratory values obtained within 30 days prior to entry:

  * Absolute neutrophil count (ANC) >=750 cells/mm^3
  * Hemoglobin >= 7.4 g/dL
  * Platelet count >= 50,000/mm^3
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=3 X upper limit of normal (ULN)
  * Total bilirubin <=2.5 X ULN
* HIV infection status must be documented as either absent or present, as defined below:

Absence of HIV-1 infection within 30 days prior to Step 2 entry OR HIV-1 infection at any time prior to Step 2 entry.

* For HIV-positive candidates only: CD4+ cell count of >=50 cells/mm^3, performed within 7 days prior to entry at a DAIDS-approved laboratory
* For females of reproductive potential, negative serum or urine pregnancy test within 7 days prior to entry. Female participants who are participating in sexual activity that could lead to pregnancy must agree to use one reliable non-hormonal method of contraception (condoms or an IUD), or another method (diaphragm or cervical cap) if it is approved by the national regulatory authority and used according to package insert, while receiving study medications.
* Willingness to be hospitalized for a minimum of 9 consecutive days.
* Ability to produce an overnight sputum sample of sufficient quality and quantity.

Exclusion Criteria for Step 1:

-There are no exclusion criteria for Step 1.

Exclusion Criteria for Step 2:

-Current treatment with INH or receipt of INH during the 7 days prior to Step 2 entry.

NOTE: Participants who have been started on INH-containing anti-TB treatment and have received this treatment for less than or equal to 2 weeks, but for whom TB drugs have been discontinued because of resistance to INH (with or without resistance to RIF), can participate in the study, but may need to be hospitalized, at the discretion of the investigator, while these drugs wash out; the minimum washout period for these drugs is 7 days.

* Protocol versions 1.0 and 2.0 only: Any prior history of treatment for MDR-TB with second-line anti-TB drugs. This includes all drugs with anti-TB activity, except INH, RIF, ethambutol, pyrazinamide, and streptomycin.
* Protocol versions 1.0 and 2.0 only: Receipt of more than 7 cumulative days of antibiotics intended for bacterial treatment that may have anti-TB activity, including amoxicillin/clavulanate (Augmentin), linezolid, metronidazole, or drugs from the quinolone class, with any of those days falling within the 14 days prior to Step 1 screening sputum collection.
* Protocol version 3.0 only: Receipt of more than 7 cumulative days of second-line anti-TB drugs (including all drugs with anti-TB activity, except INH, RIF, ethambutol, pyrazinamide, and streptomycin) and/or antibiotics intended for bacterial treatment that may have anti-TB activity, including amoxicillin/clavulanate (Augmentin), linezolid, metronidazole, or drugs from the quinolone class, with any of those days falling within the 14 days prior to Step 1 screening sputum collection. The minimum washout period for these drugs is 7 days prior to Step 2 pre-entry sputum collection.
* Known exposure to a person diagnosed with extensively drug-resistant (XDR)-TB or known personal diagnosis of XDR-TB in the past.
* Protocol version 1.0: For HIV+ participants only: Current treatment, or treatment within 30 days prior to entry, with antiretroviral therapy (ART) or expected to initiate ART within 8 days after Step 2 entry. Prior receipt of ART for the prevention of mother-to-child-transmission is not exclusionary.
* Breastfeeding.
* Known allergy/sensitivity to INH.
* Karnofsky score <60 or poor general condition where any delay in full TB treatment cannot be tolerated in the opinion of the investigator (at screening).
* Any of the following co-morbidities, complications, or underlying medical conditions:

  * Known current neurological TB (eg, TB of the spine, TB meningitis)
  * Peripheral neuropathy >=Grade 2 within 14 days prior to entry
  * Current or history of epilepsy, defined as seizure disorder requiring current treatment with an antiepileptic medicine or history of any seizures within the prior year
* Any condition as determined by physical examination, medical history, laboratory data, or chest x-ray which, in the opinion of the investigator, would interfere with participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas H Diacon, MD, PhD, Study Chair — TASK Clinical Research Center CRS, Karl Bremer Hospital; Kelly Dooley, MD, PhD, Study Chair — Johns Hopkins Adult AIDS CRS
Locations (2):
- GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS (31730), Port-au-Prince, Haiti
- TASK Applied Science CRS (31718), Bellville, South Africa

REFERENCES:
- [Derived] Gausi K, Ignatius EH, De Jager V, Upton C, Kim S, McKhann A, Moran L, Wiesner L, von Groote-Bidlingmaier F, Marzinek P, Vanker N, Yvetot J, Pierre S, Rosenkranz SL, Swindells S, Diacon AH, Nuermberger EL, Denti P, Dooley KE. High-Dose Isoniazid Lacks EARLY Bactericidal Activity against Isoniazid-resistant Tuberculosis Mediated by katG Mutations: A Randomized Phase II Clinical Trial. Am J Respir Crit Care Med. 2024 Aug 1;210(3):343-351. doi: 10.1164/rccm.202311-2004OC. PMID 38564365
- [Derived] Gausi K, Ignatius EH, Sun X, Kim S, Moran L, Wiesner L, von Groote-Bidlingmaier F, Hafner R, Donahue K, Vanker N, Rosenkranz SL, Swindells S, Diacon AH, Nuermberger EL, Dooley KE, Denti P. A Semimechanistic Model of the Bactericidal Activity of High-Dose Isoniazid against Multidrug-Resistant Tuberculosis: Results from a Randomized Clinical Trial. Am J Respir Crit Care Med. 2021 Dec 1;204(11):1327-1335. doi: 10.1164/rccm.202103-0534OC. PMID 34403326
- [Derived] Dooley KE, Miyahara S, von Groote-Bidlingmaier F, Sun X, Hafner R, Rosenkranz SL, Ignatius EH, Nuermberger EL, Moran L, Donahue K, Swindells S, Vanker N, Diacon AH; A5312 Study Team. Early Bactericidal Activity of Different Isoniazid Doses for Drug-Resistant Tuberculosis (INHindsight): A Randomized, Open-Label Clinical Trial. Am J Respir Crit Care Med. 2020 Jun 1;201(11):1416-1424. doi: 10.1164/rccm.201910-1960OC. PMID 31945300
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009) — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No drug was administered under Step 1. Data collected in Step 1 determined eligibility to Step 2. Participants in Steps 1 and 2 were enrolled from August 2014 to September 2021 at 2 non-US clinical research sites.
Groups:
- Group 1: inhA Mutation: Group 1 participants had an M. tuberculosis isolate with an inhA resistance mutation
- Group 2: Neither inhA Nor katG Mutations: Group 2 participants had drug susceptible TB and harbored neither inhA nor kat G resistance mutations
- Group 3: katG Mutation: Group 3 participants had an M. tuberculosis isolate with a katG resistance mutation.
Period: Step 1: Group Identification
Arm/Group | Group 1: inhA Mutation | Group 2: Neither inhA Nor katG Mutations | Group 3: katG Mutation | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Started | 110 | 85 | 87 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 110 | 85 | 87 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 2: Arm Randomization
Arm/Group | Group 1: inhA Mutation | Group 2: Neither inhA Nor katG Mutations | Group 3: katG Mutation | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Started | 0 | 0 | 0 | 13 | 14 | 16 | 16 | 11 | 10
Completed | 0 | 0 | 0 | 13 | 14 | 15 | 16 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Step 1 Group 1: Group 1 participants had an M. tuberculosis isolate with an inhA resistance mutation. This group only includes participants who did not proceed to step 2.
- Step 1 Group 2: Group 2 participants had drug susceptible TB and harbored neither inhA nor kat G resistance mutations. This group only includes participants who did not proceed to step 2.
- Step 1 Group 3: Group 3 participants had an M. tuberculosis isolate with a katG resistance mutation. This group only includes participants who did not proceed to step 2.
- Total: Total of all reporting groups
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort | Step 1 Group 1 | Step 1 Group 2 | Step 1 Group 3 | Total
Number analyzed (Participants) | 13 | 14 | 16 | 16 | 11 | 10 | 67 | 69 | 66 | 282
Age, Continuous [Median (Full Range); unit: years] | 31 [20 to 58] | 32 [20 to 58] | 34 [18 to 55] | 30 [19 to 58] | 36 [23 to 61] | 39 [20 to 54] | 36 [19 to 59] | 32 [18 to 63] | 35 [18 to 62] | 35 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 4 | 3 | 3 | 26 | 27 | 22 | 97
  Male | 10 | 11 | 10 | 12 | 8 | 7 | 41 | 42 | 44 | 185
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Black Non-Hispanic | 13 | 14 | 16 | 15 | 10 | 10 | 66 | 69 | 66 | 279
Region of Enrollment [Count of Participants; unit: Participants]
  Haiti | 0 | 0 | 0 | 0 | 7 | 5 | 0 | 0 | 2 | 14
  South Africa | 13 | 14 | 16 | 16 | 4 | 5 | 67 | 69 | 64 | 268
Karnofsky Score [Median (Full Range); unit: units on a scale] — Karnofsky Score measures a person's ability to perform activities of daily living. The scores range from 0 to 100, with a higher score indicating that a person is better able to perform daily activities. Population: Karnofsky Score was only collected for participants who were randomized to start study treatment.
  units on a scale
    number analyzed (Participants) | 13 | 14 | 16 | 16 | 11 | 10 | 0 | 0 | 0 | 80
    (all) | 90 [70 to 90] | 90 [70 to 90] | 80 [70 to 90] | 90 [80 to 90] | 80 [70 to 90] | 90 [80 to 90] |  |  |  | 90 [70 to 90]
BMI [Median (Full Range); unit: kg/m^2] — Population: BMI was only collected on participants who were randomized to start study treatment.
  kg/m^2
    number analyzed (Participants) | 13 | 14 | 16 | 16 | 11 | 10 | 0 | 0 | 0 | 80
    (all) | 18.1 [16.2 to 30.9] | 17.7 [14.6 to 23.6] | 18.5 [15.4 to 30.1] | 18.0 [15.2 to 29.7] | 19.3 [16.0 to 24.4] | 17.6 [14.5 to 24.3] |  |  |  | 18.1 [14.5 to 30.9]
HIV Status [Count of Participants; unit: Participants] — Population: HIV status was only collected on participants who were randomized to start study treatment.
  Participants
    Living without HIV: number analyzed (Participants) | 13 | 14 | 16 | 16 | 11 | 10 | 0 | 0 | 0 | 80
    Living without HIV | 11 | 11 | 12 | 13 | 9 | 8 |  |  |  | 64
    Living with HIV: number analyzed (Participants) | 13 | 14 | 16 | 16 | 11 | 10 | 0 | 0 | 0 | 80
    Living with HIV | 2 | 3 | 4 | 3 | 2 | 2 |  |  |  | 16

OUTCOME MEASURES:

1. Primary Outcome: Daily Change in log10 Colony-forming Unit (CFU)
Description: Negative daily change in log10 CFU indicate decreases in bacterial burden over the 7 day period. Defined as EBA0-7(CFU) = [Day 7 log10 CFU per mL - baseline log10 CFU per mL]/7. The baseline measure is the mean of the pre-entry visit and entry visit sputum colony counts.
Time Frame: Measured at baseline and Day 7
Population: Participants who took at least one dose of study treatment in Step 2 in Groups 1 and 2. CFU was not collected for Group 3. Participants who had missing Baseline or Day 7 CFU counts were not included.
Measure: Mean (Standard Deviation); unit: log10 CFU per mL sputum per day
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort
Number analyzed (Participants) | 12 | 11 | 12 | 11
log10 CFU per mL sputum per day | -0.06 (0.14) | -0.18 (0.12) | -0.21 (0.15) | -0.15 (0.11)

2. Primary Outcome: Daily Change in Time to Positivity (TTP)
Description: The time to positivity (TTP) measures growth of mycobacterium tuberculosis using MGIT assay in hours. Higher values of daily change in TTP indicate greater decrease in bacterial burden over the 7 day period and is therefore better.
  Daily change is defined as EBA0-7(TTP) = [Day 7 TTP - Baseline TTP]/7. Baseline is the mean of the pre-entry visit and entry visit TTPs.
Time Frame: Measured at baseline and Day 7
Population: Participants who took at least one dose of study treatment in Step 2. Participants who had missing Baseline or Day 7 TTP counts were not included.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 13 | 14 | 14 | 16 | 10 | 10
hours per day | 3 (8) | 8 (6) | 10 (8) | 10 (4) | 2.0 (7.9) | 4.6 (7.9)

3. Primary Outcome: INH PK Parameter Area Under the Concentration Time Curve (AUC 0-24 Hours)
Description: AUC 0-24h defines area under the concentration-time curve over the period of 24 hours post-dose, estimated through non-compartmental methods using the linear trapezoidal rule.
Time Frame: Intensive INH PK samples collected on Day 6 of INH initiation at sample times pre-dose, 0.5h, 1h, 2h, 4h, 6h, 8h, 12h and 24h post-dose.
Population: Participants in each treatment dose arm with intensive PK results in Step 2.
Measure: Median (Inter-Quartile Range); unit: ug*hr/mL
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 13 | 14 | 15 | 16 | 11 | 10
ug*hr/mL | 14.05 [9.27 to 28.73] | 53.08 [23.65 to 67.26] | 50.24 [42.24 to 89.71] | 10.47 [8.04 to 18.09] | 54.13 [37.86 to 92.57] | 70.54 [66.39 to 89.64]

4. Primary Outcome: Number of Participants With Grade 2 or Higher Drug-related Adverse Clinical or Laboratory Events
Description: Post-entry, all new diagnoses, signs/symptoms and laboratory events of ≥Grade 2 that were assessed by the site as drug related. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used.
Time Frame: Measured from entry through Day 21
Population: Participants who took at least one dose of study treatment in Step 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 13 | 14 | 16 | 16 | 11 | 10
Participants | 0 | 4 | 0 | 1 | 1 | 0

5. Secondary Outcome: INH PK Parameter Minimum Plasma Concentration (Cmin)
Description: Cmin defines minimum concentration observed over the 24 hours of the INH dosing interval.
Time Frame: as for outcome 3
Population: Participants in each treatment dose arm with intensive PK results in Step 2.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 13 | 14 | 15 | 16 | 11 | 10
ug/mL | 0.053 [0.053 to 0.053] | 0.053 [0.053 to 0.179] | 0.053 [0.053 to 0.099] | 0.053 [0.053 to 0.053] | 0.053 [0.053 to 0.329] | 0.053 [0.053 to 0.221]

6. Secondary Outcome: INH PK Parameter Maximum Plasma Concentration (Cmax)
Description: Cmax defines maximum concentration observed over the 24 hours of the INH dosing interval.
Time Frame: as for outcome 3
Population: Participants in each treatment dose arm with intensive PK results in Step 2.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 13 | 14 | 15 | 16 | 11 | 10
ug/mL | 5.26 [4.41 to 7.13] | 10.4 [8.26 to 11.90] | 15.1 [12.30 to 17.90] | 4.55 [3.62 to 6.00] | 15 [13.05 to 20.10] | 22.15 [18.10 to 23.75]

7. Secondary Outcome: INH Minimum Inhibitory Concentration (MIC) Against M. Tuberculosis Isolates
Description: MIC are determined by phenotypic drug susceptibility testing (DST) based on spot sputum collected at Step 1 Day 0. For group 3 participants shown, MIC was tested using Thermofisher Sensititre MYCOTB plates.
Time Frame: Day 0
Population: Step 1 participants in Group 3 for whom MIC results were available and tested using Thermofisher Sensititre MYCOTB plates. MIC was not done using Thermofisher Sensititre MYCOTB plates for participants enrolled under versions 1.0 and 2.0 of the protocol (including all Group 1 and 2 participants and many Group 3 participants). Three Group 3 Version 3 participants had missing MIC results. Note: Participants were not yet randomized to a treatment in Step 1 so all Group 3 participants are combined.
Measure: Count of Participants; unit: Participants
Groups:
- Step 1 Group 3 Version 3: Group 3 participants who had an M. tuberculosis strain with a katG mutation with or without an inhA mutation. This group includes all participants in Group 3 enrolled in Step 1 of the study under Version 3 of the protocol (which assessed MIC by Thermofisher MYCOTB Sensititre plate).
Arm/Group | Step 1 Group 3 Version 3
Number analyzed (Participants) | 18
Participants
  0.03 μg/mL | 1
  0.06 μg/mL | 0
  0.12 μg/mL | 0
  0.25 μg/mL | 0
  0.5 μg/mL | 0
  1 μg/mL | 1
  2 μg/mL | 4
  4 μg/mL | 9
  >4 μg/mL | 3

8. Secondary Outcome: Proportions of Participants Estimated to Have a Drop in log10 CFU/mL at or Above 0.65 log10 CFU/mL.
Description: Proportions of participants obtained through simulation using the estimated model who have a drop in log10 CFU/mL at or above the threshold of 0.65 log10 CFU/mL; 0.65 is half the drop in log10 CFU/mL observed in participants with DS-TB (Group 2) on day 7. A total of 10000 simulated pseudo-participants per arm were used based on data from the study participants. The NAT2 genotype distribution was based only on Group 1 and 2 participants since NAT2 genotype data was not available for Group 3. The simulations were run repeatedly. The point estimate of the proportion was based on the median proportion of the pseudo-individuals across the repeated simulations and the 90% confidence interval used the 5th and 95th percentiles of the proportion across the repeated simulations.
Time Frame: From baseline through day 7
Population: Data from all participants were included in the modeling.
Measure: Median (90% Confidence Interval); unit: proportion of simulated participants
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 13 | 14 | 16 | 16 | 11 | 10
proportion of simulated participants | 0.17 [0.00 to 0.60] | 0.50 [0.06 to 0.84] | 0.64 [0.18 to 0.91] | 0.88 [0.78 to 0.99] | 0.01 [0.00 to 0.30] | 0.05 [0.00 to 0.41]

9. Secondary Outcome: Daily Change in log10 CFU Measured by Early- (EBA0-2) and Late-phase (EBA2-7) Individual-based Parameter Estimates From Nonlinear Models
Description: Negative daily change in log10 CFU indicate decreases in bacterial burden over the time period. The mean CFU are estimated using all values by fitting a biphasic regression models for each participant. The daily change for the first two days of treatment was calculated as EBA0-2 (CFU)= [Day 2 log10 CFU per mL - baseline log10 CFU per mL]/2. The daily change from day 2 to day 7 was calculated as EBA2-7 (CFU)= [Day 7 log10 CFU per mL - Day 2 log10 CFU per mL]/5. Baseline is the average of pre-entry and entry visits.
Time Frame: At baseline, day 2, and day 7
Population: Four participants were excluded from the analysis due to missing CFU values in Group 1-INH 10 mg (2), Group 1-INH 15mg (1), and Group 2 (1). CFU was not collected for Group 3.
Measure: Mean (Standard Deviation); unit: log10 CFU per mL sputum per day
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort
Number analyzed (Participants) | 13 | 12 | 15 | 15
log10 CFU per mL sputum per day
  EBA(0-2) | -0.23 (0.30) | -0.17 (0.22) | -0.13 (0.39) | -0.41 (0.33)
  EBA(2-7) | -0.01 (0.15) | -0.17 (0.13) | -0.25 (0.17) | -0.07 (0.19)

10. Secondary Outcome: Daily Change in TTP Measured by Early- (EBA0-2) and Late-phase (EBA2-7) Individual-based Parameter Estimates From Nonlinear Models
Description: The time to positivity (TTP) measures growth of mycobacterium tuberculosis using MGIT assay in hours. Higher values of daily change in TTP indicate greater decrease in bacterial burden over the time period and is therefore better. The mean log transformed TTP are estimated using all values by fitting a biphasic regression models for each participant. The daily change over the first two days of treatment is calculated as EBA0-2 (TTP)= [Day 2 TTP - baseline TTP]/2. The daily change from Day 2 to Day 7 is calculated as EBA2-7 (TTP)= [Day 7 TTP - Day 2 TTP]/5. Baseline is the average of pre-evaluation and entry visits.
Time Frame: At baseline, day 2, and day 7
Population: All available TTP results were used.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 13 | 13 | 16 | 16 | 11 | 10
hours per day
  EBA(0-2) | 7.78 (17.22) | 11.03 (6.40) | 7.35 (14.73) | 22.39 (11.44) | 2.91 (3.57) | -1.36 (7.59)
  EBA(2-7) | 1.77 (9.61) | 5.45 (7.39) | 12.01 (8.29) | 5.09 (6.43) | 2.69 (12.21) | 5.45 (8.36)

11. Secondary Outcome: EBA Measured by Individual-based Parameter Estimates From Linear or Nonlinear Models When the Number of Phases Differs Between Every Dosing Cohort
Description: Both TTPs and log10 CFU from the pre-evaluation and entry visits averaged and treated as the baseline TTP and log10 CFU for each participant. This outcome was included for analysis if the number of phases differed between every dosing cohort. Since the number of phases did not differ between dosing cohorts, this outcome was not measured.
Time Frame: From baseline through day 7
Population: This outcome was not measured.
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Mean EBA Measured by Ratio of the Following Areas: Numerator = AUC of Observed log10 CFU Over 7 Days and Denominator = Baseline log10 CFU for Every Dosing Cohort in Groups 1 and 2
Description: This approach utilizes the area between baseline CFU per mL and the CFU curve for each participant, as measured using the trapezoidal rule. This outcome was included for analysis if the number of phases differed between every dosing cohort. Since the number of phases did not differ between dosing cohorts, this outcome was not measured.
Time Frame: From baseline through day 7
Population: This outcome was not measured.
Arm/Group | Group 1: 5mg Cohort | Group 1: 10mg Cohort | Group 1: 15mg Cohort | Group 2: 5mg Cohort | Group 3: 15mg Cohort | Group 3: 20mg Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Measured from baseline through Day 21
Description: For participants who took at least one dose of study treatment in Step 2, all new diagnoses (per ACTG criteria for clinical events and other diseases), signs/symptoms (S/S) of grade 2 or higher or any S/S that led to a change in treatment regardless of grade, and all laboratory events regardless of grade. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used. Adverse events were only collected on participants who started study treatment. No treatment was administered in Step 1.
Groups:
- Group 1- INH 5mg: Group 1 participants had an M. tuberculosis strain with an inhA mutation only. 5 mg cohort received Isoniazid 5 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
- Group 1- INH 10mg: Group 1 participants had an M. tuberculosis strain with an inhA mutation only. 10 mg cohort received Isoniazid 10 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
- Group 1- INH 15mg: Group 1 participants had an M. tuberculosis strain with an inhA mutation only. 15 mg cohort received Isoniazid 15 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
- Group 2- INH 5mg: Group 2 participants had an M. tuberculosis strain with neither inhA nor katG mutations. All Group 2 participants received Isoniazid 5 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
- Group 3- INH 15mg: Group 3 participants had an M. tuberculosis strain with a katG mutation with or without an inhA mutation. 15mg cohort received Isoniazid 15 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
- Group 3- INH 20mg: Group 3 participants had an M. tuberculosis strain with a katG mutation with or without an inhA mutation. 20mg cohort received Isoniazid 20 mg/kg daily plus vitamin B6 >=25 mg daily for 7 days
Arm/Group | Group 1- INH 5mg | Group 1- INH 10mg | Group 1- INH 15mg | Group 2- INH 5mg | Group 3- INH 15mg | Group 3- INH 20mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/16 | 0/16 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/14 | 0/16 | 1/16 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 12/13 | 14/14 | 15/16 | 16/16 | 11/11 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1- INH 5mg (N=13) | Group 1- INH 10mg (N=14) | Group 1- INH 15mg (N=16) | Group 2- INH 5mg (N=16) | Group 3- INH 15mg (N=11) | Group 3- INH 20mg (N=10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1- INH 5mg (N=13) | Group 1- INH 10mg (N=14) | Group 1- INH 15mg (N=16) | Group 2- INH 5mg (N=16) | Group 3- INH 15mg (N=11) | Group 3- INH 20mg (N=10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tuberculous pleurisy (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3 | 5 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 4 | 4 | 0 | 1
Blood albumin (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 11 | 14 | 15 | 16 | 11 | 10
Blood alkaline phosphatase increased (Investigations) | 1 | 3 | 4 | 1 | 0 | 3
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 4 | 6 | 5 | 4 | 6 | 4
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Informed Consent Form (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT01936831/Prot_ICF_000.pdf
  • Statistical Analysis Plan: Primary Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT01936831/SAP_001.pdf
  • Statistical Analysis Plan: Pharmacology Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT01936831/SAP_002.pdf